CLINICAL TRIAL: NCT01448746
Title: Optimal Prophylactic Method of Venous Thromboembolism for Gastrectomy in Korean Patients
Brief Title: Optimal Prophylactic Method of Venous Thromboembolism (VTE)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Kyo Young Song, Associate Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CUMC-GC2011
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Venous Thromboembolism
Keywords: gastric cancer; VTE; incidence
MeSH Terms: conditions — Venous Thromboembolism; Stomach Neoplasms | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intermittent pneumatic compression (Experimental): another arm include intermittent pneumatic compression plus low molecular weight heparin
  Interventions: Drug: low molecular weight heparin

INTERVENTIONS:
Drug: low molecular weight heparin — 40mg 12 hours before surgery and 12 hours later surgery

SUMMARY:
This study is to define the optimal method of prophylaxis for patients with gastrectomy in Korea and the investigators hypothesized only mechanical method would be enough for preventing VTE on perioperative period.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is common and often fatal complication in patients with cancer.

Gastric cancer is the most frequent cancer in Korea.

The incidence of VTE would be increased in patients with gastric cancer, especially associated surgery.

However, the incidence and optimal prophylactic method associated with cancer surgery are not well studied in Asian patients.

Most Korean surgeon concerns regarding the increased postoperative bleeding associated with low molecular weight heparin(LMWH)prophylaxis.

The incidence and adverse event will be examined to define the optimal prophylactic method of VTE in surgical patients with gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as gastric cancer
* Elective and curative under general anesthesia
* ECOG score 0-2
* ASA score 3 or less than 3
* Informed consents

Exclusion Criteria:

* 2nd primary cancer
* VTE history within one year
* Anticoagulation history
* Allergic to heparin
* Pregnancy or expected pregnancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2011-10; Primary Completion 2016-01 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
incidence of VTE | up to 30 days after operation
  The incidence of VTE between mechanical method only group and mechnical plus LMWH group.

SECONDARY OUTCOMES:
Adverse event | up to 30 days after operation
  The adverse event such as bleeding will also be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Kyo Young Song, M.D., Principal Investigator — The Catholic University of Korea
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kakkos S, Kirkilesis G, Caprini JA, Geroulakos G, Nicolaides A, Stansby G, Reddy DJ. Combined intermittent pneumatic leg compression and pharmacological prophylaxis for prevention of venous thromboembolism. Cochrane Database Syst Rev. 2022 Jan 28;1(1):CD005258. doi: 10.1002/14651858.CD005258.pub4. PMID 35089599
- [Derived] Kahale LA, Matar CF, Hakoum MB, Tsolakian IG, Yosuico VE, Terrenato I, Sperati F, Barba M, Schunemann H, Akl EA. Anticoagulation for the initial treatment of venous thromboembolism in people with cancer. Cochrane Database Syst Rev. 2021 Dec 8;12(12):CD006649. doi: 10.1002/14651858.CD006649.pub8. PMID 34878173
- [Derived] Kahale LA, Matar CF, Tsolakian I, Hakoum MB, Barba M, Yosuico VE, Terrenato I, Sperati F, Schunemann H, Akl EA. Oral anticoagulation in people with cancer who have no therapeutic or prophylactic indication for anticoagulation. Cochrane Database Syst Rev. 2021 Oct 8;10(10):CD006466. doi: 10.1002/14651858.CD006466.pub7. PMID 34622445
- [Derived] Jung YJ, Seo HS, Park CH, Jeon HM, Kim JI, Yim HW, Song KY. Venous Thromboembolism Incidence and Prophylaxis Use After Gastrectomy Among Korean Patients With Gastric Adenocarcinoma: The PROTECTOR Randomized Clinical Trial. JAMA Surg. 2018 Oct 1;153(10):939-946. doi: 10.1001/jamasurg.2018.2081. PMID 30027281
- [Derived] Song KY, Yoo HM, Kim EY, Kim JI, Yim HW, Jeon HM, Park CH. Optimal prophylactic method of venous thromboembolism for gastrectomy in Korean patients: an interim analysis of prospective randomized trial. Ann Surg Oncol. 2014 Dec;21(13):4232-8. doi: 10.1245/s10434-014-3893-1. Epub 2014 Jul 11. PMID 25012265